CLINICAL TRIAL: NCT06007300
Title: A Multiomics Study Based on the Dynamic Evolution of Endometrial Carcinogenesis
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY-2023-136-B
Record Dates: First submitted 2023-08-09; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: the Dynamic Evolution of Endometrial Carcinogenesis; Multiomics Analysis
Keywords: Dynamic Evolution; Genomics; Transcriptome; Proteomics; Metabolomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal Group: Patients with normal endometrium
- Precancerous Group: Patients with atypical hyperplasia of endometrium
- Carcinoma Group: Patients with endometrial cancer

SUMMARY:
The goal of this observational study is to draw the characteristic maps of imaging omics, genomics, transcriptome, proteomics, pathological omics, metabolomics, etc. of the dynamic evolution of endometrial carcinogenesis in 100 patients with normal endometrium, 100 patients with atypical endometrial hyperplasia, and 100 patients with endometrial cancer; and then to explore the underlying molecular mechanism, and establish the database system for the dynamic evolution of endometrial carcinogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis: normal endometrium, atypical hyperplasia endometrium, or endometrial cancer;
* Obtain pathological results after undergoing hysteroscopic surgery or hysterectomy;
* The patient voluntarily participated in this research project with good compliance and was able to complete the enrollment according to the experimental requirements;
* Sign the informed consent form and consent to the collection and use of their data, and consent to genomics, transcriptome and other tests.

Exclusion Criteria:

* Patients with malignant tumors in other parts of the body;
* Suffering from uncontrollable neurological diseases, psychiatric diseases, or psychiatric disorders;
* Poor compliance and inability to cooperate and describe treatment responders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with normal endometrium (requiring diagnostic or therapeutic hysteroscopy or hysterectomy for other reasons), patients with precancerous lesions of endometrium, and patients with endometrial cancer who underwent surgery in the gynecology and obstetrics department of Renji Hospital affiliated to Shanghai Jiaotong University School of Medicine, whose illness was diagnosed as normal endometrium, atypical hyperplasia endometrium, or endometrial cancer by pathology.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
The mutant genes of participants and their expression as assessed by gene sequencing, RNA sequencing and mass spectrometry analysis | August 2023 to June 2026
Differences in the expression of these mutant genes among the three groups of participants as assessed by SAS® 9.4 | January 2026 to June 2026